CLINICAL TRIAL: NCT05793385
Title: The Uncommon Complications of Meckel's Diverticulum: a Single Center Case Series Study and Literature Review
Brief Title: The Uncommon Complications of Meckel's Diverticulum
Acronym: MD
Status: Completed | Type: Observational
Sponsor: Haramaya Unversity (Other)
Responsible Party: Principal Investigator, Badhaasaa, Assistant professor, Haramaya Unversity
Other Study IDs: HU/31/10/2022
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: To Report the Rare Occurrence of Meckel's Diverticulum
Keywords: Meckel's diverticulum; isolated torsion; intussusception; acute abdomen; acute appendicitis
MeSH Terms: conditions — Meckel Diverticulum; Intussusception; Abdomen, Acute; Appendicitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: operative intervention — all patients were operated after being admitted to surgical ward for acute abdomen

SUMMARY:
Acas series study was conducted on emergency acute abdomen patients who finally confirmed intraoperatively as Meckel's diverticulum with different complications. Simple perforation to isolated axial torsioned gangrene was observed. The patients signed consent for their cases to be published.

DETAILED DESCRIPTION:
The study was aimed at reporting the rare complications of Meckel's diverticulum, which were diagnosed intraoperatively among acute abdomen patients presented to HFCSH. The patients had different complications ranging from simple isolated perforation to gangrenous Meckel's diverticulum. All of the patients gave their informed written and signed consent for publication.

ELIGIBILITY:
Inclusion Criteria:

* all patients diagnosed with complicated meckel's diverticulum

Exclusion Criteria:

* patients who didn't consent

Ages: 4 Years to 33 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients who presented with the diagnosis of acute abdomen
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Outcome upon discharge | 10 months
  outcome of patients with different complications were reported even though there was no death.

CONTACTS AND LOCATIONS:
Locations (1):
- Haramaya university, Harar, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Its against our institutions rule and regulations to share patient data to the third party